CLINICAL TRIAL: NCT04930497
Title: Immediate Implant Placement Using Vestibular Socket Therapy With and Without Bone Grafting (Randomized Controlled Clinical Trial)
Brief Title: Vestibular Socket Therapy With and Without Bone Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VST_bone grafting
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Tooth Extraction
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vestibular socket technique with bone grafting (Experimental)
  Interventions: Procedure: vestibular socket technique with bone grafting
- vestibular socket technique without bone grafting (Active Comparator)
  Interventions: Procedure: vestibular socket technique without bone grafting

INTERVENTIONS:
Procedure: vestibular socket technique with bone grafting — a vestibular horizontal incision was made then a subperiosteal tunnel was created and a facial bone membrane was placed. The facial gap was filled with a mixture of autogenous bone and deproteinized bovine bone mineral
  Arms: vestibular socket technique with bone grafting
Procedure: vestibular socket technique without bone grafting — the vestibular incision was done horizontally about 3 to 4 mm apical to the mucogingival junction and extending 5 to 10 mm horizontally. A submucoperiosteal tunnel was created labially from the socket orifice till the vestibular access incision
  Arms: vestibular socket technique without bone grafting

SUMMARY:
Management of the jumping gap in the Vestibular Socket Therapy. And to study what is the best technique to manage this gap for optimal esthetic result.

DETAILED DESCRIPTION:
22 patients were randomly assigned to Group 1: Had received implants with the vestibular socket technique accompanied with bone grafting the jumping gap between the implant and the labial membrane.

Group 2: Had received implants with the vestibular socket technique, but without bone grafting the jumping gap.

Facial bone thickness and height were evaluated using CBCT scans at baseline before tooth extraction and after 6 and 13 months

ELIGIBILITY:
Inclusion Criteria:

* presence of a hopeless tooth or teeth in the esthetic zone (maxillary anterior area)
* No active infection
* Adequate bone palatally and apically
* Presence of contralateral tooth for the tooth being replaced

Exclusion Criteria:

* Hopeless tooth with acute infection
* heavy smokers (more than 10 cigarettes per day)
* pregnant and patients received recent chemotherapy/radiotherapy (during the previous year)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Facial bone thickness | baseline, 6 months and 13 months
  using CBCT scans (Carestream 8000D, Carestream Dental)
Change in Facial bone height | baseline, 6 months and 13 months
  using CBCT scans (Carestream 8000D, Carestream Dental)

CONTACTS AND LOCATIONS:
Locations (1):
- Private Practice Clinic, Alexandria, Egypt